CLINICAL TRIAL: NCT04451070
Title: Impact of Clinic First Curricular Transformation on Family Medicine Resident Burnout at an Air Force Family Medicine Residency
Brief Title: Impact of Curricular Transformation on Family Medicine Resident Burnout
Status: Completed | Type: Observational
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: FWH20200114E
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Burnout Among Family Medicine Resident Physicians
Keywords: Burnout; Family Medicine; Resident; Clinic First
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Family Medicine resident physicians: Family Medicine resident physicians at David Grant Medical Center who started their Family Medicine residency at David Grant Medical Center between June 2018 - June 2019 and are scheduled to graduate from Family Medicine residency between June 2021 - June 2022.
  Interventions: Other: Clinic First curriculum

INTERVENTIONS:
Other: Clinic First curriculum — The Clinic First model was designed by the Association of Family Medicine Residency Directors (AFMRD) in collaboration with the University of California San Francisco's (UCSF) Center for Excellence in Primary Care. The components of the Clinic First model are summarized in the Association of American Medical Colleges' (AAMC) publication titled "High-Functioning Primary Care Residency Clinics: Building Blocks for Providing Excellent Care and Training". Using the principles of Clinic First, the authors of this study drafted a Family Medicine residency curriculum to be implemented at David Grant Medical Center at the beginning of the 2020-2021 academic year.

SUMMARY:
The purpose of this study is to determine if the implementation of a Family Medicine residency curriculum that is based upon the principles of Clinic First, as originally described by the Center for Excellence in Primary Care at the University of California, San Francisco, results in a decrease in the extent of burnout among Family Medicine resident physicians at David Grant Medical Center on Travis Air Force Base in Fairfield, California.

This is a descriptive study designed to assess the extent of burnout among Family Medicine resident physicians pre- and post-implementation of a Clinic First-inspired Family Medicine residency curriculum. The study will utilize the Maslach Burnout Inventory Human Services Survey for Medical Personnel (MBI-HSS (MP)), which is a validated instrument that was designed to assess (1) emotional exhaustion, (2) depersonalization, and (3) personal accomplishment among medical personnel.

DETAILED DESCRIPTION:
This is a descriptive study designed to assess the extent of burnout among Family Medicine resident physicians pre- and post-implementation of a Clinic First-inspired Family Medicine residency curriculum. The study will utilize the Maslach Burnout Inventory Human Services Survey for Medical Personnel (MBI-HSS (MP)). The MBI-HSS (MP) is a validated instrument that was designed to assess (1) emotional exhaustion, (2) depersonalization, and (3) personal accomplishment among medical personnel. The survey will be administered anonymously as a series of 3 surveys both prior to and following the implementation of a Clinic-First inspired curriculum.

Survey Period #1: Baseline - within 3 months prior to Clinic First implementation Survey Period #2: Short Term - 3-6 months after Clinic First implementation Survey Period #3: Intermediate Term - 9-12 months after Clinic First implementation

The MBI-HSS (MP) will be administered anonymously using printed paper copies to all eligible Family Medicine resident physicians who are in attendance at a Family Medicine residency didactics session within the respective survey period. An independent support staff member from the Clinical Investigations Facility (CIF) will introduce the research study to the resident physicians in attendance using a uniform script and administer the surveys. All Family Medicine resident physicians who meet the eligibility criteria and who are in attendance on the designated didactics day will be provided with a paper copy of the MBI-HSS (MP) and given ample time to complete the questionnaire. The eligible respondents will also be given a separate demographic questionnaire that was generated by the researchers and collects information on gender, age, ethnicity, and marital status. The completed surveys and demographic questionnaires will be collected by the CIF support staff member and de-identified using a using a 4 digit numerical code generated from randomizer.org. The code will be used to link future surveys that are answered by the same resident physician.

For those resident physicians who are not in attendance at the designated didactics session, paper copies of the survey and demographic questionnaire will be placed in their personal mailboxes. An email (email address provided by investigators) will be sent to those resident physicians from a member of the CIF support staff informing them that they have 2 weeks to complete the survey and demographic questionnaire and instructing them to place completed surveys/questionnaires in a labeled manila envelope next to the personal mailboxes. The CIF support staff member will pick-up the labeled manila envelope at the end of the 2 week period and de-identify the surveys as described above. This process will be repeated for each survey period such that each eligible resident physician will complete 3 surveys. The MBI-HSS (MP) will be administered as similarly as possible for all participants both pre- and post-curricular transformation to avoid confounding factors.

Responses to survey questions will be entered into an Excel spreadsheet by the CIF support staff to be readied for the statistician. Responses will be given numerical data values for analysis. Since all of the questions in the MBI-HSS (MP) have already been assigned numerical value, the responses will be coded accordingly. Descriptive statistics (e.g. frequencies and percentages) will be used to for analysis. For each participant, the level of burnout for each sub-section will be calculated using the MBI scoring results/interpretation, and will be compared across the three time points (ie, baseline, 3-6 months following implementation, and 9-12 months after implementation).

Demographic information will be collected to describe the sample.

The investigators acknowledge that there may be missing data if resident physicians decline to complete the MBI-HSS (MP), decline to answer all of the questions within the MBI-HSS (MP), or fail to answer subsequent surveys after completing the baseline MBI-HSS (MP). A response rate for each question within each survey period will be calculated and reported. Incomplete surveys will still be reviewed and included in the final data.

All analyses will be performed using STATA v.13.0 (College Station, TX).

ELIGIBILITY:
Inclusion Criteria:

* Family Medicine resident physicians at David Grant Medical Center
* Residents must have started their Family Medicine residency at David Grant Medical Center between June 2018 - June 2019
* Residents must be scheduled to graduate from Family Medicine residency between June 2021 - June 2022

Exclusion Criteria:

* Family Medicine resident physicians at David Grant Medical Center who started their residency before June 2018 or after June 2019.
* Family Medicine resident physicians at David Grant Medical Center who are scheduled to graduate from Family Medicine residency before May 2021 or after July 2022.

Ages: 25 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: Family Medicine resident physicians in the Family Medicine residency program at David Grant Medical Center on Travis Air Force Base in Fairfield, California who fulfill the eligibility criteria as listed above.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Family Medicine resident physician burnout, baseline | Baseline (before new curriculum was implemented)
  Family Medicine resident physician burnout as measured by the Maslach Burnout Inventory Human Services Survey for Medical Personnel (MBI-HSS-MP). Participants will rate how often they experience each of the 22 symptom questions on a scale of 0 (never) to 6 (every day). Both a total score and an average score for each of the 3 subscales (ie, emotional exhaustion, depersonalization, and personal accomplishments) will be calculated.
Family Medicine resident physician burnout, 3-6 months | 3-6 months after new curriculum was implemented
  Family Medicine resident physician burnout as measured by the Maslach Burnout Inventory Human Services Survey for Medical Personnel (MBI-HSS-MP). Participants will rate how often they experience each of the 22 symptom questions on a scale of 0 (never) to 6 (every day). Both a total score and an average score for each of the 3 subscales (ie, emotional exhaustion, depersonalization, and personal accomplishments) will be calculated.
Family Medicine resident physician burnout, 9-12 months | 9-12 months after new curriculum was implemented
  Family Medicine resident physician burnout as measured by the Maslach Burnout Inventory Human Services Survey for Medical Personnel (MBI-HSS-MP). Participants will rate how often they experience each of the 22 symptom questions on a scale of 0 (never) to 6 (every day). Both a total score and an average score for each of the 3 subscales (ie, emotional exhaustion, depersonalization, and personal accomplishments) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney E Halista, MD, Principal Investigator — Family Medicine Faculty Physician at David Grant Medical Center; Heather A Dalton, MD, Principal Investigator — Family Medicine Faculty Physician at David Grant Medical Center
Locations (1):
- David Grant Medical Center, Fairfield, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Accreditation Council for Graduate Medical Education. "The ACGME Releases 'CLER National Report of Findings 2019: Initial Visits to Sponsoring Institutions With 2 or Fewer Core Residency Programs'." PR Newswire: Press Release Distribution, Targeting, Monitoring and Marketing, Accreditation Council for Graduate Medical Education, 22 Aug. 2019, www.prnewswire.com/newsreleases/the-acgme-releases-cler-national-report-of-findings-2019-initial-visits-to-sponsoringinstitutions-with-2-or-fewer-core-residency-programs-300905975.html.
- [Background] 2. Wagner, Robin. David Grant Medical Center Clinical Learning Environment Review (CLER) Site Visit Report. Accreditation Council for Graduate Medical Education, 2019, pp. 1-21, David Grant Medical Center Clinical Learning Environment Review (CLER) Site Visit Report.
- [Background] 3. "ACGME Program Requirements for Graduate Medical Education in Family Medicine." Accreditation Council for Graduate Medical Education , 1 July 2019, www.msm.edu/Education/GME/Documents/FamilyMedicine/ACGME_Requirements_120_family_medicine_2016.pdf.
- [Background] 4. Bodenheimer, Thomas, et al. High-Functioning Primary Care Residency Clinics: Building Blocks for Providing Excellent Care and Training. Association of American Medical Colleges, 2016, pp. 1-62, High-Functioning Primary Care Residency Clinics: Building Blocks for Providing Excellent Care and Training.
- [Background] 5. "Clinic First Collaborative." Association of Family Medicine Residency Directors (AFMRD), 2020, www.afmrd.org/page/afmrdmembership.
- [Background] Wallace JE, Lemaire JB, Ghali WA. Physician wellness: a missing quality indicator. Lancet. 2009 Nov 14;374(9702):1714-21. doi: 10.1016/S0140-6736(09)61424-0. PMID 19914516
- [Background] 7. "Burn-out an 'Occupational Phenomenon': International Classification of Diseases." World Health Organization, World Health Organization, 28 May 2019, www.who.int/mental_health/evidence/burn-out/en/.
- [Background] Dupras DM, West CP. Training for Careers in Primary Care: Time for Attention to Culture. J Gen Intern Med. 2015 Sep;30(9):1243-4. doi: 10.1007/s11606-015-3416-1. No abstract available. PMID 26173533
- [Background] 9. Shapiro, Miriam, and Alice Fornari. Factors Influencing Primary Care Residency Selection among Students at an Urban Private Medical School. 1st ed., vol. 25, The Einstein Journal of Biology and Medicine, 2010, pp. 19-24, Factors Influencing Primary Care Residency Selection among Students at an Urban Private Medical School.
- [Background] Alavi M, Ho T, Stisher C, Richardson E, Kelly C, McCrory K, Snellings J, Zurek K, Boltz MW. Factors That Influence Student Choice in Family Medicine A National Focus Group. Fam Med. 2019 Feb;51(2):143-148. doi: 10.22454/FamMed.2019.927833. PMID 30736039